CLINICAL TRIAL: NCT00006361
Title: A Phase II Trial of SU5416 (NSC #696819) in Patients With Advanced or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: SU5416 in Treating Patients With Advanced or Recurrent Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068232; MSKCC-00049; NCI-79
Record Dates: First submitted 2000-10-04; First posted 2003-05-30 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2002-12

CONDITIONS: Carcinoma of Unknown Primary; Head and Neck Cancer; Non-melanomatous Skin Cancer
Keywords: squamous cell carcinoma of the skin; recurrent skin cancer; stage IV nasopharyngeal cancer; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; squamous cell carcinoma of unknown primary; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary; Head and Neck Neoplasms; Skin Neoplasms; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Semaxinib

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of cancer cells by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of SU5416 in treating patients who have advanced or recurrent cancer of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of SU5416 on survival and tumor response in patients with advanced or recurrent squamous cell carcinoma of the head and neck.
* Determine the safety and toxicity of SU5416 in these patients.

OUTLINE: Patients receive SU5416 IV over 1 hour twice weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed for 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within 1.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven epidermoid/squamous cell carcinoma of the oral cavity, lip, hypopharynx, oropharynx, nasopharynx, sinonasal tract, or larynx; undifferentiated carcinoma of the nasopharynx (WHO type III); sinonasal undifferentiated carcinoma; or squamous cell carcinoma of unknown primary or the skin with initial presentation in the head and neck region
* Advanced or recurrent disease that is incurable with surgery or radiotherapy
* No more than 2 prior cytotoxic chemotherapy regimens for recurrent, persistent, or metastatic disease

  * Prior exposure to chemopreventive agents (e.g., tretinoin or other vitamin analogues) is not considered to be a prior cytotoxic chemotherapy exposure
* At least 1 measurable indicator lesion

  * Bone metastases, elevated enzyme levels, or lesions on radionuclide scans are not acceptable as the sole parameters of measurable disease
* No history of brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Hemoglobin greater than 8 g/dL
* Platelet count greater than 100,000/mm3
* No history of coagulation disorder

Hepatic:

* Bilirubin normal
* SGOT less than 2.5 times upper limit of normal
* PT no greater than 14 seconds
* aPTT no greater than 40 seconds

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncompensated coronary artery disease
* No myocardial infarction or severe/unstable angina within the past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No deep venous or arterial thrombosis within the past 3 months
* No unstable cardiac rhythm
* No cerebrovascular accident within the past 6 months

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* No history of allergic reaction to paclitaxel
* No other active malignancy except:

  * Basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Synchronous epidermoid/squamous cell carcinoma of the head and neck (oral cavity, lip, hypopharynx, oropharynx, nasopharynx, sinonasal tract, or larynx)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active bacterial infection requiring antibiotics
* No other concurrent medical condition that would increase risk

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Pfister, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Zahalsky AJ, Wong RJ, Lis E, et al.: Phase II trial of SU5416 in patients with advanced incurable head and neck cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-902, 2002.